CLINICAL TRIAL: NCT01997918
Title: Haploidentical Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) in the Treatment of Relapse After a First Allogeneic HSCT: a Retrospective Cohort Study by the German Cooperative Transplant Study Group
Brief Title: Secondary Haplo HSCT for Relapse After Initial Allogeneic HSCT
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); University Hospital Augsburg (Other)
Responsible Party: Sponsor
Other Study IDs: KTS 2. Haplo HSCT
Record Dates: First submitted 2013-10-29; First posted 2013-11-28 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Relapse of Hematological Malignancies
Keywords: Secondary allogeneic HSCT; Haploidentical HSCT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Relapse of underlying hematologic malignancies after allogeneic hematopoietic stem cell transplantation (HSCT) is frequently treated by a second allogeneic HSCT (HSCT2). Choosing an alternative donor is often advocated to maximize chances of a graft versus tumour (GVT) effect. We and others published that success of this strategy when using an alternative human leukocyte antigen (HLA) identical donor is limited, at least when acute leukemia is the underlying disease. The aggressivity of the rapidly proliferating leukemia seems to prevail over GVT effects. A more potent alloimmune response is observed following haploidentical HSCT, especially early after haploidentical HSCT. This might be related to a fast and large expansion of natural killer (NK)-cells. Their alloreactive effect might translate into higher rates of tumor control. On the other hand, non-relapse complications (treatment related mortality, TRM) might be high in advanced relapsed tumour patients with heavy pretreatment and due to delayed immune reconstitution after haploidentical HSCT. The use of a haploidentical donor for HSCT2 following a first allogeneic HSCT from an HLA identical donor has been so far only systematically evaluated in small retrospective single center reports. Thus, in this multicenter study we aim to collect data on the extent to which participating centers employ haploidentical transplantation in the situation of relapse after HSCT2.

DETAILED DESCRIPTION:
Relapse of underlying hematologic malignancies after allogeneic hematopoietic stem cell transplantation (HSCT) is frequently treated by a second allogeneic HSCT (HSCT2). Choosing an alternative donor is often advocated to maximize chances of a graft versus tumour (GVT) effect. We and others published that success of this strategy when using an alternative HLA identical donor is limited, at least when acute leukemia is the underlying disease. The aggressivity of the rapidly proliferating leukemia seems to prevail over GVT effects. A more potent alloimmune response is observed following haploidentical HSCT, especially early after haploidentical HSCT. This might be related to a fast and large expansion of NK-cells. Their alloreactive effect might translate into higher rates of tumor control. On the other hand, non-relapse complications (treatment related mortality, TRM) might be high in advanced relapsed tumour patients with heavy pretreatment and due to delayed immune reconstitution after haploidentical HSCT. The use of a haploidentical donor for HSCT2 following a first allogeneic HSCT from an HLA identical donor has been so far only systematically evaluated in small retrospective single center reports. Thus, in this multicenter study we aim to collect data on the extent to which participating centers employ haploidentical transplantation in the situation of relapse after HSCT2. We will describe and quantify the specific patient, donor, treatment, graft and outcomes characteristics associated with the course of treatment. To assess and control for the bias that is associated with the retrospective nature of this study, we will emphasize to collect clearly stated reasons for the decision to use a haploidentical transplant, e.g. as opposed to drug therapy or a second transplant from the original or an alternative HLA identical donor. This is a retrospective observational cohort study. German centers performing allogeneic HSCT are asked to contribute. Data will be validated and missing information will be further retrieved by the four principal investigators through phone. Final follow up will be performed in April 2014, 2014. To be able to supply durable data on the primary endpoints, only patients receiving a haploidentical HSCT2 between 01.07.2003 and 30.06.2013 will be included.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years at time of HSCT2
* Malignant hematologic disease
* Informed consent signed by the patients on the use of data in registry analyses
* 1st allogeneic HSCT performed from any donor, including haploidentical HSCT1
* Hematological or extramedullary relapse after HSCT1
* Haploidentical 2nd allogeneic HSCT (i.e. >= 2 Antigen mismatch family donor) between 01.07.2003 and 30.06.2013

Third or higher allogeneic HSCT does not preclude analysis as long as HSCT2 was haploidentical.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving salvage secondary haploidentical allogeneic HSCT after failure of primary allogeneic HSCT
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Treatment related mortality (TRM) of haploidentical HSCT2 | up to day 365
Toxicity of haploidentical HSCT2 | up to day 365
  NCI Common Terminology Criteria for Adverse Events (CTCAE) v.4

SECONDARY OUTCOMES:
complete remission (CR) rate after haploidentical HSCT2 | day 100
Overall survival (OS) at 2 years after haploidentical HSCT2 | 2 years
Graft versus host disease (GVHD) after haploidentical HSCT2 | 2 years
Incidence of rejection after haploidentical HSCT2 | 1 year
Disease free survival (DFS) at 2 years after haploidentical HSCT2 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang A Bethge, MD, Principal Investigator — University Hospital Tuebingen; Christoph Schmid, MD, Principal Investigator — University Hospital Augsburg; Johanna Tischer, MD, Principal Investigator — Ludwig-Maximilians University Hospital Munich; Maximilian Christopeit, MD, Principal Investigator — University Hospital of Halle